CLINICAL TRIAL: NCT00931164
Title: Single-center Phase I/II Trial of Sodium Oxybate in Patients With Alternating Hemiplegia of Childhood (AHC-SO Trial)
Brief Title: Sodium Oxybate in Patients With Alternating Hemiplegia of Childhood (AHC-SO)
Acronym: AHC-SO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Alternating Hemiplegia of Childhood Foundation (Other); Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Kathryn Swoboda, Associate Professor, Neurology and Pediatrics Director, Pediatric Motor Disorders Research Program, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32164; 103932
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Alternating Hemiplegia of Childhood
Keywords: phase I/II study; effects of sodium oxybate; cohort of 6 children and young adults; AHC
MeSH Terms: conditions — Alternating hemiplegia of childhood | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium oxybate (Experimental): * The study is an open-label, Phase I/II trial designed to obtain additional safety and pharmacokinetic parameters for use of sodium oxybate in children and adolescents afflicted with AHC.
  * Given the limited number of children carrying the diagnosis of AHC, typical controls will not be available for our study. In lieu of this, the subjective recording of ictal episodes in the 6 week period prior to drug initiation will serve as reference in determining drug efficacy.
  Interventions: Drug: Sodium Oxybate

INTERVENTIONS:
Drug: Sodium Oxybate — dosage is by weight

SUMMARY:
WHO: The investigators are recruiting children and young adults to participate in a research study who:

1. Have been diagnosed with Alternating Hemiplegia of Childhood (AHC)
2. Are between the ages of 6 months - 25 years old
3. Have at least three 10-minute-long AHC episodes during a typical week
4. Can commit to 12 weeks of completing of a daily log describing AHC episodes and to a multi-night hospital stay at the University of Utah Center for Clinical and Translational Science (CCTS)

WHY: The goal of this study is to evaluate whether the study drug can safely and effectively decrease AHC episodes and improve the quality of life of individuals with AHC.

WHAT and WHERE: This study involves at least 12 weeks of completing and submitting daily AHC Episode Logs and a five-day hospital stay at the University of Utah CCTS.

There are 4 phases of the study, and they include:

1. Six weeks of daily log completion prior to starting study drug
2. Five day stay at the University of Utah CCTS
3. Six additional weeks of daily log completion while using study drug at home
4. One day clinic visit to the University of Utah for follow up

COMPENSATION:

There is no fee to participate. All procedures performed specifically for this study will be covered by the study and will not be billed to you or your insurance company.

The study drug will be dispensed to you free of charge. Meals and lodging at the study site will be provided free of charge for the study participant and one care provider. Additionally, the research team will assist subjects with booking and obtaining free transportation, such as an airline tickets, to and from the study site.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria.

* AHC classic criteria:

  * Onset of symptomatology prior to 18 months of age
  * Repeated attacks of hemiplegia involving either side of the body
  * Paroxysmal disturbances, including tonic or dystonic spells, oculomotor abnormalities, and various autonomic phenomena, during hemiplegic bouts or in isolation
  * Episodes of bilateral hemiplegia or quadriplegia starting either as generalization of a hemiplegic episode or bilateral from the beginning
  * Immediate disappearance of symptoms upon sleeping, with possible resumption 10-20 minutes after waking
  * Evidence of developmental delay and neurologic abnormalities including choreoathetosis, dystonia, or ataxia

In addition:

* Provision of a complete daily event log for 6 weeks prior to initiation of sodium oxybate therapy, including the: (1) frequency, (2) duration, (3) type, (4) severity of episodes, and (5) therapies, if any, used in an attempt to abort the episode
* Ages 6 months to 25 years at the time of study enrollment
* Minimum of 3 AHC episodes weekly, lasting at least 10 minutes each, on average prior to study enrollment
* Brain neuroimaging studies excluding alternative etiology for symptoms
* Documented absence of epileptiform features on EEG during typical ictal events
* Ability of primary caregivers of study participants to submit online daily AHC Episode Logs indicating frequency and duration of ictal episodes over the entire study period
* Written informed consent from parents/guardians and assent from children 7 years or older
* Girls/women > 12 years of age will be required to be on birth control continuously if they are considered at risk to become pregnant. Those not on birth control will be required to have a screening pregnancy test at baseline, and to confirm their willingness to practice birth control or abstain from sexual activity for the duration of treatment with study medication.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation.

* History of hepatic insufficiency, renal insufficiency, significant respiratory disease, cardiac arrhythmia, congenital heart defect, hypertension, or ischemic stroke
* History of allergy/sensitivity to sodium oxybate
* Use of sodium oxybate within 30 days of study enrollment
* Serious illness requiring systemic treatment and/or hospitalization within two weeks prior to study enrollment
* Change in neurologic medication regimen within 30 days of study enrollment.
* Inability to stay at the Center for Clinical and Translational Science (CCTS) for 5 days due to behavioral issues
* Unwillingness or inability to travel to study site during the necessary 1 week titration period to determine the most appropriate dose of GHB for subsequent administration
* Noncompliance with AHC Episode Log or study visit requirements
* Sleep apnea not adequately treated with C-PAP and oxygen saturation monitoring prior to drug therapy initiation
* Succinic semialdehyde dehydrogenase deficiency

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J. Swoboda, M.D., Principal Investigator — University of Utah/Primary Children's Medical Center
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Addolorato G, Cibin M, Capristo E, Beghe F, Gessa G, Stefanini GF, Gasbarrini G. Maintaining abstinence from alcohol with gamma-hydroxybutyric acid. Lancet. 1998 Jan 3;351(9095):38. doi: 10.1016/s0140-6736(05)78088-0. No abstract available. PMID 9433435
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Background] Arnold DL, Silver K, Andermann F. Evidence for mitochondrial dysfunction in patients with alternating hemiplegia of childhood. Ann Neurol. 1993 Jun;33(6):604-7. doi: 10.1002/ana.410330608. PMID 8498840
- [Background] Bourgeois M, Aicardi J, Goutieres F. Alternating hemiplegia of childhood. J Pediatr. 1993 May;122(5 Pt 1):673-9. doi: 10.1016/s0022-3476(06)80003-x. PMID 8496742
- [Background] Bourgeois M, Aicardi J. The treatment of alternating hemiplegia of childhood with flunarizine: experience with 17 patients. Alternating Hemiplegia of Childhood, edited by F Andermann, J Aicardi, and F Vigevano. 1995;191-194.
- [Background] Caputo F, Addolorato G, Stoppo M, Francini S, Vignoli T, Lorenzini F, Del Re A, Comaschi C, Andreone P, Trevisani F, Bernardi M; Alcohol Treatment Study Group. Comparing and combining gamma-hydroxybutyric acid (GHB) and naltrexone in maintaining abstinence from alcohol: an open randomised comparative study. Eur Neuropsychopharmacol. 2007 Dec;17(12):781-9. doi: 10.1016/j.euroneuro.2007.04.008. Epub 2007 Jul 3. PMID 17611081
- [Background] Casaer P. Flunarizine in alternating hemiplegia in childhood. An international study in 12 children. Neuropediatrics. 1987 Nov;18(4):191-5. doi: 10.1055/s-2008-1052478. PMID 3320807
- [Background] Casaer P, Azou M. Flunarizine in alternating hemiplegia in childhood. Lancet. 1984 Sep 8;2(8402):579. doi: 10.1016/s0140-6736(84)90794-3. No abstract available. PMID 6147627
- [Background] Defossez M, Le Bec G, Sancier A, Manelfe C, Espagno MT, Bouzat A, Sevely A. [Neuro-sedation and cranial C.-T. scan in infants and children (author's transl)]. Anesth Analg (Paris). 1979;36(11-12):525-9. French. PMID 554477
- [Background] Ferrara SD, Giorgetti R, Zancaner S, Orlando R, Tagliabracci A, Cavarzeran F, Palatini P. Effects of single dose of gamma-hydroxybutyric acid and lorazepam on psychomotor performance and subjective feelings in healthy volunteers. Eur J Clin Pharmacol. 1999 Jan;54(11):821-7. doi: 10.1007/s002280050560. PMID 10027654
- [Background] Frucht SJ, Bordelon Y, Houghton WH, Reardan D. A pilot tolerability and efficacy trial of sodium oxybate in ethanol-responsive movement disorders. Mov Disord. 2005 Oct;20(10):1330-7. doi: 10.1002/mds.20605. PMID 15986420
- [Background] Haan J, Kors EE, Terwindt GM, Vermeulen FL, Vergouwe MN, van den Maagdenberg AM, Gill DS, Pascual J, Ophoff RA, Frants RR, Ferrari. Alternating hemiplegia of childhood: no mutations in the familial hemiplegic migraine CACNA1A gene. Cephalalgia. 2000 Oct;20(8):696-700. doi: 10.1046/j.0333-1024.2000.00095.x. PMID 11167897
- [Background] Hunter AS, Long WJ, Ryrie CG. An evaluation of gamma-hydroxybutyric acid in paediatric practice. Br J Anaesth. 1971 Jun;43(6):620-8. doi: 10.1093/bja/43.6.620. No abstract available. PMID 5089942
- [Background] Jiang W, Chi Z, Ma L, Du B, Shang W, Guo H, Wu W. Topiramate: a new agent for patients with alternating hemiplegia of childhood. Neuropediatrics. 2006 Aug;37(4):229-33. doi: 10.1055/s-2006-924721. PMID 17177149
- [Background] Jen J, Yue Q, Nelson SF, Yu H, Litt M, Nutt J, Baloh RW. A novel nonsense mutation in CACNA1A causes episodic ataxia and hemiplegia. Neurology. 1999 Jul 13;53(1):34-7. doi: 10.1212/wnl.53.1.34. PMID 10408533
- [Background] Kanavakis E, Xaidara A, Papathanasiou-Klontza D, Papadimitriou A, Velentza S, Youroukos S. Alternating hemiplegia of childhood: a syndrome inherited with an autosomal dominant trait. Dev Med Child Neurol. 2003 Dec;45(12):833-6. doi: 10.1017/s0012162203001543. PMID 14667076
- [Background] Katchan B, Mamelak M, Hwang P. Alternating Hemiplegia of Childhood: Rationale for the use of Gammahydroxybutyrate, Reprints from the 10th International Child Neurology Congress, Montreal, June 2006.
- [Background] Kemp GJ, Taylor DJ, Barnes PR, Wilson J, Radda GK. Skeletal muscle mitochondrial dysfunction in alternating hemiplegia of childhood. Ann Neurol. 1995 Oct;38(4):681-4. doi: 10.1002/ana.410380421. PMID 7574469
- [Background] Kothare SV, Adams R, Valencia I, Faerber EC, Grant ML. Improved sleep and neurocognitive functions in a child with thalamic lesions on sodium oxybate. Neurology. 2007 Apr 3;68(14):1157-8. doi: 10.1212/01.wnl.0000258658.00692.36. No abstract available. PMID 17404202
- [Background] Kyriakides T, Drousiotou A. No structural or biochemical evidence for mitochondrial cytopathy in a case of alternating hemiplegia of childhood. Ann Neurol. 1994 Nov;36(5):805-6. doi: 10.1002/ana.410360529. No abstract available. PMID 7979233
- [Background] Mamelak M, Black J, Montplaisir J, Ristanovic R. A pilot study on the effects of sodium oxybate on sleep architecture and daytime alertness in narcolepsy. Sleep. 2004 Nov 1;27(7):1327-34. doi: 10.1093/sleep/27.7.1327. PMID 15586785
- [Background] Meyer S, Gottschling S, Georg T, Lothschutz D, Graf N, Sitzmann FC. Gamma-hydroxybutyrate versus chlorprothixene/phenobarbital sedation in children undergoing MRI studies. Klin Padiatr. 2003 Mar-Apr;215(2):69-73. doi: 10.1055/s-2003-38500. PMID 12677545
- [Background] Micieli G, Sances G, Pacchetti C, Trucco M, Magri M, Piazza D. Flunarizine: a wide spectrum prophylactic for migraine headache. Int J Clin Pharmacol Res. 1984;4(3):239-45. PMID 6490242
- [Background] Mikati M. Alternating hemiplegia of childhood. Pediatr Neurol. 1999 Oct;21(4):764. doi: 10.1016/s0887-8994(99)00090-9. No abstract available. PMID 10580894
- [Background] Mikati MA, Kramer U, Zupanc ML, Shanahan RJ. Alternating hemiplegia of childhood: clinical manifestations and long-term outcome. Pediatr Neurol. 2000 Aug;23(2):134-41. doi: 10.1016/s0887-8994(00)00157-0. PMID 11020638
- [Background] Murali H, Kotagal S. Off-label treatment of severe childhood narcolepsy-cataplexy with sodium oxybate. Sleep. 2006 Aug;29(8):1025-9. doi: 10.1093/sleep/29.8.1025. PMID 16944670
- [Background] Nimmerrichter AA, Walter H, Gutierrez-Lobos KE, Lesch OM. Double-blind controlled trial of gamma-hydroxybutyrate and clomethiazole in the treatment of alcohol withdrawal. Alcohol Alcohol. 2002 Jan-Feb;37(1):67-73. doi: 10.1093/alcalc/37.1.67. PMID 11825860
- [Background] Poschl J, Kolker S, Bast T, Brussau J, Ruef P, Linderkamp O, Bettendorf M. Gamma-hydroxybutyric acid sedation in neonates and children undergoing MR imaging. Klin Padiatr. 2007 Jul-Aug;219(4):217-9. doi: 10.1055/s-2007-973056. PMID 17638167
- [Background] Priori A, Bertolasi L, Pesenti A, Cappellari A, Barbieri S. gamma-hydroxybutyric acid for alcohol-sensitive myoclonus with dystonia. Neurology. 2000 Apr 25;54(8):1706. doi: 10.1212/wnl.54.8.1706. No abstract available. PMID 10762526
- [Background] Ricci S. Sleep studies of children with alternating hemiplegia of childhood. Alternating Hemiplegia of Childhood, edited by Andermann, Aicardi, and Vigevano. 1995;95-98.
- [Background] Rinalduzzi S, Valeriani M, Vigevano F. Brainstem dysfunction in alternating hemiplegia of childhood: a neurophysiological study. Cephalalgia. 2006 May;26(5):511-9. doi: 10.1111/j.1468-2982.2006.01066.x. PMID 16674759
- [Background] Scrima L, Hartman PG, Johnson FH Jr, Thomas EE, Hiller FC. The effects of gamma-hydroxybutyrate on the sleep of narcolepsy patients: a double-blind study. Sleep. 1990 Dec;13(6):479-90. doi: 10.1093/sleep/13.6.479. PMID 2281247
- [Background] Sasaki M, Sakuragawa N, Osawa M. Long-term effect of flunarizine on patients with alternating hemiplegia of childhood in Japan. Brain Dev. 2001 Aug;23(5):303-5. doi: 10.1016/s0387-7604(01)00229-7. PMID 11504600
- [Background] Silver K, Andermann F. Alternating hemiplegia of childhood: a study of 10 patients and results of flunarizine treatment. Neurology. 1993 Jan;43(1):36-41. doi: 10.1212/wnl.43.1_part_1.36. PMID 8423908
- [Background] Silver K, Andermann F. Alternating hemiplegia of childhood: treatment with flunarizine. Alternating Hemiplegia of Childhood, edited by F Andermann, J Aicardi, and F Vigevano. 1995;195-198.
- [Background] Suner S, Szlatenyi CS, Wang RY. Pediatric gamma hydroxybutyrate intoxication. Acad Emerg Med. 1997 Nov;4(11):1041-5. doi: 10.1111/j.1553-2712.1997.tb03677.x. PMID 9383489
- [Background] Swoboda KJ, Kanavakis E, Xaidara A, Johnson JE, Leppert MF, Schlesinger-Massart MB, Ptacek LJ, Silver K, Youroukos S. Alternating hemiplegia of childhood or familial hemiplegic migraine? A novel ATP1A2 mutation. Ann Neurol. 2004 Jun;55(6):884-7. doi: 10.1002/ana.20134. PMID 15174025
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860
- [Background] U.S. Xyrem Multicenter Study Group. Sodium oxybate demonstrates long-term efficacy for the treatment of cataplexy in patients with narcolepsy. Sleep Med. 2004 Mar;5(2):119-23. doi: 10.1016/j.sleep.2003.11.002. PMID 15033130
- [Background] Verret S, Steele JC. Alternating hemiplegia in childhood: a report of eight patients with complicated migraine beginning in infancy. Pediatrics. 1971 Apr;47(4):675-80. No abstract available. PMID 5089756
- [Background] Weaver TE, Cuellar N. A randomized trial evaluating the effectiveness of sodium oxybate therapy on quality of life in narcolepsy. Sleep. 2006 Sep;29(9):1189-94. doi: 10.1093/sleep/29.9.1189. PMID 17040006
- [Background] Xyrem International Study Group. A double-blind, placebo-controlled study demonstrates sodium oxybate is effective for the treatment of excessive daytime sleepiness in narcolepsy. J Clin Sleep Med. 2005 Oct 15;1(4):391-7. PMID 17564408
- [Background] Xyrem International Study Group. Further evidence supporting the use of sodium oxybate for the treatment of cataplexy: a double-blind, placebo-controlled study in 228 patients. Sleep Med. 2005 Sep;6(5):415-21. doi: 10.1016/j.sleep.2005.03.010. PMID 16099718

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Oxybate: * The study is an open-label, Phase I/II trial designed to obtain additional safety and pharmacokinetic parameters for use of sodium oxybate in children and adolescents afflicted with AHC.
  * Given the limited number of children carrying the diagnosis of AHC, typical controls will not be available for our study. In lieu of this, the subjective recording of ictal episodes in the 6 week period prior to drug initiation will serve as reference in determining drug efficacy.
  Sodium Oxybate : dosage is by weight
Period: Overall Study
Arm/Group | Sodium Oxybate
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.4 [1.1 to 11.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5
  Ireland | 1

OUTCOME MEASURES:

1. Primary Outcome: Time Duration of AHC Episodes
Time Frame: Week 7
Reporting Status: Not Posted

2. Primary Outcome: Observed Safety Data During 5-day Hospitalization for Drug Dose Identification
Time Frame: Week 7
Reporting Status: Not Posted

3. Primary Outcome: Number of Participants Who Reported Side Effects During Home Drug Maintenance Phase
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 6
participants | 4

4. Secondary Outcome: Mean Daily Percentage of Time That Functional Status is Affected Due to Episodes
Time Frame: Week 14
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life Questionnaires
Time Frame: Week 14
Reporting Status: Not Posted

6. Secondary Outcome: Mood and Behavior Questionnaires
Time Frame: Week 14
Reporting Status: Not Posted

7. Secondary Outcome: Functional Skills Questionnaires
Time Frame: Week 14
Reporting Status: Not Posted

8. Secondary Outcome: Neuropsychological Tests
Time Frame: Week 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sodium Oxybate
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate (N=6)
Loss of consciousness/vomit event (Gastrointestinal disorders) | 1 (2)
Respiratory Distress Event (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate (N=6)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Otitis Media (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Heat Rash (General disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes